CLINICAL TRIAL: NCT01924000
Title: Minoxidil 1% for Eyebrow Enhancement: A Randomized , Double-blind , Placebo-controlled , Split-face Comparative Study
Brief Title: Minoxidil 1% for Eyebrow Enhancement
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mae Fah Luang University Hospital (Other)
Responsible Party: Principal Investigator, Chuchai TANGLERTSAMPAN, MD, Instructor, Mae Fah Luang University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REH-56059
Record Dates: First submitted 2013-08-13; First posted 2013-08-16 (Estimated); Last update posted 2014-04-22 (Estimated); Status verified 2014-04

CONDITIONS: Eyebrow Hypotrichosis; Thin Eyebrow

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Minoxidil lotion 1% (Experimental): Minoxidil lotion 1% is applied twice daily to one eyebrow.
  Interventions: Drug: Minoxidil lotion 1%
- Placebo (Placebo Comparator): Placebo is applied twice daily to the other eyebrow.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Minoxidil lotion 1% — Minoxidil lotion 1% is applied twice daily to one eyebrow.
  Arms: Minoxidil lotion 1%
Drug: Placebo
  Other Names: Placebo is applied twice daily on the other eyebrow.
  Arms: Placebo

SUMMARY:
The purpose of the study is to compare efficacy and safety of minoxidil 1% versus placebo in enhancement of eyebrows.

ELIGIBILITY:
Inclusion Criteria:

* male or female aged 18-60 years
* hypotrichosis of eyebrows
* healthy
* informed consent obtained

Exclusion Criteria:

* underlying diseases
* alopecia areata or trichotillomania
* thyroid diseases
* pregnancy or breast feeding
* previous eyebrow tattoo, trauma or accident.
* history of eyebrow or hair medications in 6 months
* history of minoxidil or its ingredient allergy
* history of eyebrow surgery.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2013-12; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
The change of global photographic assessment after 16 weeks from baseline | baseline and 16 weeks

SECONDARY OUTCOMES:
The change of hair diameter after 16 weeks from baseline | baseline and 16 weeks

OTHER OUTCOMES:
The change in number of hairs after 16 weeks from baseline | baseline and 16 weeks
Number of participants with adverse events. Adverse events include any skin rashes or symptoms. | 16 weeks
Patient satisfaction by self-assessment questionnaires | baseline and 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Chuchai Tanglertsampan, MD, Principal Investigator — Mae Fah Luang University Hospital (Bangkok)
Locations (1):
- Mae Fah Luang University Hospital (Bangkok), Bangkok, Thailand

REFERENCES:
- [Result] Suwanchatchai W, Tanglertsampan C, Pengsalae N, Makornwattana M. Efficacy and safety of bimatoprost 0.03% versus minoxidil 3% in enhancement of eyebrows: a randomized, double-blind, split-face comparative study. J Dermatol. 2012 Oct;39(10):865-6. doi: 10.1111/j.1346-8138.2012.01579.x. Epub 2012 May 17. No abstract available. PMID 22594928
- See also: Related Info — http://www.mfu.ac.th/2012eng/